CLINICAL TRIAL: NCT06902623
Title: A Phase II Study of Treatment De-Escalation for Favorable Prognosis, Stage I-II Human Papilloma Virus (HPV) or p16-Positive Oropharyngeal Cancer Receiving Definitive Radiotherapy
Brief Title: Treatment De-Escalation for Favorable Prognosis Human Papilloma Virus (HPV) or p16-Positive Oropharyngeal Cancer Receiving Definitive Radiotherapy
Acronym: Lombardi197
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000197
Record Dates: First submitted 2025-03-03; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Oropharyngeal Cancers; HPV; Tonsil Cancer; Base of Tongue Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms; Tonsillar Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Radiation only (Experimental): Radiation therapy only to a dose of 66Gy to gross disease
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiation only to 66Gy

SUMMARY:
The current standard treatment option for Human Papillomavirus (HPV) or p16-positive oropharyngeal cancer is full-dose radiation combined with chemotherapy. Results with chemotherapy combined with full-dose radiation therapy leads to high rates of cure; this has called into question whether therapy can be decreased in intensity since both chemotherapy and radiation have long-term side effects. One approach to decrease intensity of treatment is to give radiation alone (excluding chemotherapy) and to decrease radiation therapy dose. The investigator believes that omitting chemotherapy and decreasing radiation dose both to tumor and the regions of the head and neck at highest risk of potential spread, may have no significant impact on the cancer recurring while potentially leading to fewer long-term side effects.

DETAILED DESCRIPTION:
This study aims to estimate the efficacy of radiation dose de-escalation while omitting chemotherapy for favorable prognosis HPV or p16-positive oropharyngeal cancer patients receiving definitive radiation therapy, where efficacy is measured by 2-year progression free survival (PFS) rate after treatment de-escalation for low-risk HPV+ oropharyngeal squamous cell carcinoma. This study also aims to determine quality of life parameters, complete clinical and radiographic response, as well as local, regional and distant metastasis control as well as overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age on the day of signing informed consent.
* Patients must have a diagnosis of p16+ and/or HPV+ squamous cell carcinoma of the oropharynx (including base of tongue, glossotonsilar sulcus, tonsil, soft palate, vallecula, and/or posterior oropharyngeal wall).
* clinical stage stage I-II (T1-2 N1 M0, or T3 N0-1 M0 ) (AJCC 8th ed.) SCCA of the oropharynx that would mandate definitive chemoradiation as current standard of care when standard radiation fractionation is applied. Debulking of the disease by resecting the exophytic portion of the tumor for biopsy/sample or symptom alleviation will be permitted, as long as gross unresected tumor is left behind.
* Subjects must agree to biopsy of areas that are FDG-avid on PET-CT scan 3-4 months after treatment.
* Patients must have Karnofsky Performance Status (KPS) ≥ 60 within 8 weeks prior to registration
* Patients must have had a neutrophil:lymphocyte ratio ≤ 5 within 8 weeks of registration.
* Patient must have had a hemoglobin count ≥ 10 within 8 weeks of registration. The patient may receive transfusion to reach this goal.
* Patients must be a current non-smoker (at least 6 months) with ≤ 15 pack-year smoking history
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients with gross involvement of level 4 lymph node level
* Endophytic T3 disease, as clinically determined by the principal investigator.
* Patients with any single lymph node > 4cm (multiple lymph nodes including nodal conglomerates that in sum measure >4cm is allowed)
* Patients with nodal disease clinically fixed to or radiographically invading adjacent neck musculature any single lymph node > 4cm (multiple lymph nodes including nodal conglomerates that in sum measure >4cm is allowed)
* Prior history of malignancy diagnosed within 2 years prior to registration, except for nonmelanomatous skin cancer that has completed treatment and the patient is deemed as being disease-free, or Gleason 6 prostate cancer undergoing active surveillance.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Progression Free Survival- 2-year progression free survival, as determined by standard of care physical examination and standard of care surveillance imaging.

SECONDARY OUTCOMES:
Local Control of disease (LC) rate | 2 years
  Number of patient with local control at 2 years, as determined by standard of care physical examination and/or standard of care surveillance imaging.
Regional Control of diseaes (RC) rate | 2 years
  Number of patient with regional control at 2 years, as determined by standard of care physical examination and/or standard of care surveillance imaging.
Distant Metastasis-Free Survival (DMFS) rate | 2 years
  Distant Metastasis-Free Survival as determined by standard of care physical examination and standard of care surveillance imaging at 2 years.
Overall Survival (OS) | 2 years
  Defined a time from start of treatment until end of study or death.
Quality of life (QOL) Core Questionnaire | 2 years
  Estimate differences in quality of life (QOL) parameters between patients treated with intensity-modulated photon radiation therapy versus proton beam radiation therapy (RT) related to radiation dose to organs at risk (OAR). QOL will be measured by validated questionnaires relating to patient related outcomes. Completed at baseline, and then at 1-2 weeks, 3 months, 6, 12, 18 and 24 months after completion of RT. EORTC QLQ Core Questionnaire (EORTC QLQ-C30), scale 0-100 with 100 being the best outcome.
Quality of life (QOL) Head and Neck Cancer | 2 years
  Estimate differences in quality of life (QOL) parameters between patients treated with intensity-modulated photon radiation therapy versus proton beam radiation therapy (RT) related to radiation dose to organs at risk (OAR). QOL will be measured by validated questionnaires relating to patient related outcomes. Completed at baseline, and then at 1-2 weeks, 3 months, 6, 12, 18 and 24 months after completion of RT. Head and Neck Cancer (QLQ-H&N35), scale 0-100 with 100 being the best outcome.
Rate of percutaneous endocsopic gastrostomy (PEG) tube placement | 1 year
  Number of patients with PEG tube placement and presence of PEG tube at 1 year in patients who are treated with de-escalated definitive radiotherapy.
Rate of neck dissection | 12 weeks post treatment completion
  Number of subjects with neck dissection within 12 weeks of treatment completion due to equivocal examination findings, even if the neck dissection shows no residual disease.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ahn, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Medstar Southern Maryland Hospital Center, Clinton, Maryland

IPD SHARING:
Plan to Share IPD: No